CLINICAL TRIAL: NCT02747251
Title: The Effects of Additional Home-based Strengthening Exercises in Shoulder Impingement Rehabilitation (The SEXSI-Trial): A Pragmatic Randomized Controlled Trial.
Brief Title: Strengthening Exercises in Shoulder Impingement (SExSI) Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Copenhagen University Hospital, Hvidovre (Other)
Collaborators: Metropolitan University College (Other); University of Copenhagen (Other); Aalborg University (Other)
Responsible Party: Principal Investigator, Mikkel Bek Clausen, PhD-Student, Copenhagen University Hospital, Hvidovre
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: H-16016763
Record Dates: First submitted 2016-04-19; First posted 2016-04-21 (Estimated); Last update posted 2020-01-23 (Actual); Status verified 2020-01

CONDITIONS: Subacromial Impingement Syndrome
Keywords: "Shoulder Impingement Syndrome"[Mesh]; "Rehabilitation"[Mesh]; "Exercise"[Mesh]; "Rotator Cuff"[Mesh]
MeSH Terms: conditions — Shoulder Impingement Syndrome

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Strengthen your Shoulder & Usual Care (Experimental): Instructions in a home-based intervention consisting of progressive high volume resistance training with an elastic band. Instructions provided 0, 2, 5, and 10 weeks after baseline. Usual care includes all treatment received by a patient during the time between baseline and follow-up, except that included in "Strengthen your Shoulder".
  Interventions: Other: Strengthen your Shoulder; Other: Usual Care
- Usual Care (Active Comparator): Includes all treatment received by a patient during the time between baseline and follow-up, except that included in "Strengthen your Shoulder".
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Strengthen your Shoulder — A simple home-based elastic band strengthening exercise intervention. This program consists of progressive high volume resistance training exercises with an elastic band.
  Arms: Strengthen your Shoulder & Usual Care
Other: Usual Care — Usual care, consisting of a referral to general rehabilitation in the municipal under the Danish Health Act § 140, most often with the alternative option to choose a private physiotherapeutic clinic, partly at their own expense. Also includes any additional treatment the patient receives between baseline and follow-up, except that included in "Strengthen your Shoulder".

SUMMARY:
This study evaluates the addition of a high dose of simple home-based elastic band strengthening exercises to usual care in patients with subacromial impingement syndrome. Half of the participants receive instructions in simple home-based elastic band strengthening exercises in addition to usual care, while the other half receive usual care.

DETAILED DESCRIPTION:
The SEXSI trial is a pragmatic, assessor and participant blinded, randomized, controlled, superiority trial, with a two-group parallel design. Patients with subacromial impingement syndrome will be randomized to either usual care or a home-based intervention consisting of progressive high volume resistance training in addition to usual care using a 1:1 allocation. The primary end-point will be change in the Shoulder Pain and Disability Index (SPADI) 16 weeks after baseline.

The overall frame for the trial is a main clinical effectiveness-part and an embedded mechanistic part. The clinical effectiveness-part will be reported in the main trial paper, and include the following outcomes: SPADI (primary outcome), Abduction strength, External rotation strength, Abduction ROM, Pain last week, QoL-index, QoL-VAS, Global impression of change and PASS. Missing outcome data will be imputed using multiple imputations based on the following variables: All previous scores in the relevant outcome, Age, Gender and Allocation.

A full trial protocol will be published and made publicly available. A constrained Linear Mixed Model (cLMM) will be applied for all continuous outcomes with Time Frame 16 weeks (including the primary outcome), to compare the change from baseline to 16 weeks in the intervention group (IG) to that in the control group (CG). The outcome at 16 weeks will be included as dependent variable, treatment group (IG or CG) as main effect and both baseline score and any additional follow up measurements as repeated measurements. The covariance structures will be selected based on the MAICE procedure. Binary outcomes will be reported as proportions with corresponding 95% confidence intervals, and will be compared using Chi-squared tests, and Odds Ratios computed from random effects logistic regression models. All of these analyses will be conducted as intention to treat (ITT) analyses, including all randomized participants, regardless of protocol adherence, meaning that all participants will be analysed as randomized. In the primary trial report, all collected outcomes will be listed, and it will be stated that the below-mentioned variables - belonging to the mechanistic part - will be reported in secondary publications.

The mechanistic part will be reported in secondary papers with a clear reference to the primary trial and trial registration, and it will hold the label "secondary analyses from a pragmatic randomized controlled trial" in the title. The following outcomes will be reported:

Outcomes regarding pain sensitization (temporal summation of pain, conditioned pain modulation, pain pressure threshold and pain catastrophizing) will be reported in a subsequent paper where we also plan to investigate:

* the modifying effects of pain sensitization on the effectiveness of the add-on intervention
* the dose-response relationship between objectively monitored adherence to the add-on intervention and change in SPADI, shoulder abduction strength and external rotation strength
* the dose-response relationship between pain sensitization and change in SPADI, shoulder abduction strength and external rotation strength, and to what degree this is mediated through adherence to the intervention.

Outcomes regarding scapula dyskinesia and scapula dysfunction will be reported in another subsequent paper, were we also plan to investigate the modifying effects of scapula dyskinesia and scapula dysfunction on the effectiveness of the intervention on changes in SPADI, abduction strength and external rotation strength.

ELIGIBILITY:
Inclusion Criteria:

* Convened for the first time to the clinic, for examination of their current shoulder disorder
* Shoulder disorder lasting at least three months
* Living in Capitol Region of Denmark
* Not pregnant
* Do not permanently use strong pain medication
* Able to understand spoken and written Danish
* ≥3 positive of the five diagnostic test for subacromial impingement syndrome (Hawkins-Kennedy test, Neer's test, pain-full arc, Resisted External Rotation test and Jobe's test)
* Offered a rehabilitation plan due to a medically justified need for general rehabilitation after discharge from the hospital under the Danish Health Act § 140.
* Completed Shoulder Pain And Disability Index (SPADI) questionnaire on the day of the medical examination

Exclusion Criteria:

* A radiologically verified new or previous fracture related to the shoulder joint, including the scapula
* Clinically suspected Glenohumeral osteoarthritis
* A clinically suspected luxation or sub-luxation of the glenohumeral, acromioclavicular or sternoclavicular joint
* A clinically suspected labral lesion, complete tear of the rotator cuff, frozen shoulder or other competing diagnoses (i.e. rheumatoid arthritis, cancer, neurological disorders, fibromyalgia, psychiatric illness)

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2016-05-13 (Actual); Primary Completion 2018-10-29 (Actual); Study Completion 2019-07 (Actual)

PRIMARY OUTCOMES:
SPADI | 16 weeks
  Shoulder Pain And Disability Index score (continuous)
  For all continuous outcomes with Time Frame 16 weeks, a constrained Linear Mixed Model (cLMM) is applied to compare the change from baseline to 16 weeks in the intervention group (IG) to that in the control group (CG), with the outcome at 16 weeks as dependent variable, treatment group (IG or CG) as main effect and both baseline score and any additional follow up measurements as repeated measurements. The covariance structures will be selected based on the MAICE procedure. These analyses will be conducted as intention to treat (ITT) analyses, including all randomized participants, regardless of protocol adherence. Participants will be analysed as randomized.

SECONDARY OUTCOMES:
Abduction strength | 16 weeks
  Maximum isometric voluntary contraction in shoulder abduction (continuous)
External rotation strength | 16 weeks
  Maximum isometric voluntary contraction in shoulder external rotation (continuous)
Abduction ROM | 16 weeks
  Active range of motion in shoulder abduction (continuous)
Pain last week | 16 weeks
  The average of least pain and average pain last week (continuous)
QoL-index | 16 weeks
  Health related Quality of Life measured using the Danish EQ-5D-3L index (continuous)
QoL-index | 52 weeks
  Health related Quality of Life measured using the Danish EQ-5D-3L index (continuous)
QoL-VAS | 16 weeks
  Health related Quality of Life measured using the Danish EQ-5D-3L VAS (continuous)
QoL-VAS | 52 weeks
  Health related Quality of Life measured using the Danish EQ-5D-3L VAS (continuous)
PCS | 16 weeks
  Pain Catastrophizing measured using the Pain Catastrophizing Scale (continuous)
Temporal summation of pain (TS) | 16 weeks
  The increase in pain recorded on an electronic VAS scale (range: 0-10 cm), during repeated standardized pressure induced pain stimuli (continuous)
CPM-Threshold | 16 weeks
  Conditioned pain threshold modulation, the percent increase in pressure pain tolerance threshold, when experimental tonic pain is induced (continuous)
CPM-Detection | 16 weeks
  Conditioned pain detection modulation, the percent increase in pressure pain detection threshold , when experimental tonic pain is induced (continuous)
PPT-deltoid | 16 weeks
  Pain pressure threshold at the deltoid muscle: The pressure applied with a manual algometer when the sensation changes from a sensation of pressure to the first sensation of pain (continuous).
PPT-Supraspinatus | 16 weeks
  Pain pressure threshold at the supraspinatus muscle: The pressure applied with a manual algometer when the sensation changes from a sensation of pressure to the first sensation of pain (continuous).
PPT-Infraspinatus | 16 weeks
  Pain pressure threshold at the infraspinatus muscle: The pressure applied with a manual algometer when the sensation changes from a sensation of pressure to the first sensation of pain (continuous).
PPT-worst | 16 weeks
  Pain pressure threshold at the site of worst pain: The pressure applied with a manual algometer when the sensation changes from a sensation of pressure to the first sensation of pain (continuous).
Sick leave | 52 weeks
  The number of days with reported sick leave due to shoulder disorder (continuous)
Global impression of change | 16 weeks
  Much improved or recovered? (Binary) Binary outcomes will be reported as proportions with corresponding 95% confidence intervals, and will be compared using a Chi-squared tests, and Odds Ratios computed from random effects logistic regression models.
PASS | 16 weeks
  Patient Acceptable Symptom State: Is the symptom state acceptable? (Binary)
Surgery | 52 weeks
  Surgery performed for the shoulder disorder? (Binary)
SDT | 16 weeks
  Scapula dyskinesia measured using the Scapula Dyskinesia Test (Binary)
mSAT | 16 weeks
  Scapula dysfunction measured using the modified Scapula Assistance Test (Binary)
SPADI | 52 weeks
  Shoulder Pain And Disability Index score (continuous)

CONTACTS AND LOCATIONS:
Overall Officials: Mikkel B Clausen, PhD-Student, Principal Investigator — Bachelor's Degree Programme in Physiotherapy, Department of Physiotherapy and Occupational Therapy, Faculty of Health and Technology, Metropolitan University College
Locations (1):
- Orthopaedic Department, Hvidovre Hospital, Hvidovre, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Clausen MB, Krohn LM, Rathleff MS, Bandholm T, Jensen SN, Christensen KB, Holmich P, Thorborg K. The Effect of Adding a Large Dose of Shoulder Strengthening to Nonoperative Care for Subacromial Impingement on Shoulder Disability, Quality of Life, Sick Days, and Surgery Rates: 1-Year Results From a Pragmatic, Double-Blind Randomized Controlled Trial (SExSI). Orthop J Sports Med. 2025 Oct 20;13(10):23259671251374314. doi: 10.1177/23259671251374314. eCollection 2025 Oct. PMID 41140544
- [Derived] Clausen MB, Rathleff MS, Graven-Nielsen T, Bandholm T, Christensen KB, Holmich P, Thorborg K. Level of pain catastrophising determines if patients with long-standing subacromial impingement benefit from more resistance exercise: predefined secondary analyses from a pragmatic randomised controlled trial (the SExSI Trial). Br J Sports Med. 2023 Jul;57(13):842-848. doi: 10.1136/bjsports-2022-106383. Epub 2023 Mar 10. PMID 36898767
- [Derived] Clausen MB, Holmich P, Rathleff M, Bandholm T, Christensen KB, Zebis MK, Thorborg K. Effectiveness of Adding a Large Dose of Shoulder Strengthening to Current Nonoperative Care for Subacromial Impingement: A Pragmatic, Double-Blind Randomized Controlled Trial (SExSI Trial). Am J Sports Med. 2021 Sep;49(11):3040-3049. doi: 10.1177/03635465211016008. Epub 2021 May 28. PMID 34048281
- [Derived] Clausen MB, Bandholm T, Rathleff MS, Christensen KB, Zebis MK, Graven-Nielsen T, Holmich P, Thorborg K. The Strengthening Exercises in Shoulder Impingement trial (The SExSI-trial) investigating the effectiveness of a simple add-on shoulder strengthening exercise programme in patients with long-lasting subacromial impingement syndrome: Study protocol for a pragmatic, assessor blinded, parallel-group, randomised, controlled trial. Trials. 2018 Mar 2;19(1):154. doi: 10.1186/s13063-018-2509-7. PMID 29499710